CLINICAL TRIAL: NCT06184490
Title: Prone Position With Different Types of Cushions in Patients With Acute Respiratory Distress Syndrome - Effects on Mechanics, Oxygenation, and Electrical Impedance Tomography Imaging
Brief Title: Prone Position With Different Types of Cushions in Patients With ARDS
Acronym: PronEIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0323
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Prone Position; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual prone position (No Intervention): Prone position with thoraco-abdominal support (cushions on the chest and hips, leaving the abdomen free)
- Modified prone position (Experimental): Prone position with lateral support (lateral cushions on the chest, hips and abdomen)
  Interventions: Procedure: Prone position with thoraco-abdominal cushion

INTERVENTIONS:
Procedure: Prone position with thoraco-abdominal cushion — Prone position with cushions positioned laterally on the chest, abdomen, and pelvis
  Arms: Modified prone position

SUMMARY:
The prone maneuver is a well-established therapy in ARDS. Traditionally, the maneuver is perform with thoraco-abdominal cushions. The goal of this study is assess, using electrical impedance tomography, whether the arrangement mode of the cushions alters lung recruitment during the prone maneuver in patients with moderate to severe ARDS.

DETAILED DESCRIPTION:
The prone position is a ventilatory therapeutic strategy used in the treatment of patients with moderate to severe Acute Respiratory Distress Syndrome (ARDS) that promotes improved oxygenation with consequent reduction in mortality. Despite being safe and effective, it is not without complications, with pressure injuries being one of the main concerns. The use of cushions helps prevent such injuries, but they can interfere with ventilatory mechanics depending on where they are placed. The aim of this study is to assess whether there is a difference in ventilatory mechanics when performing the prone maneuver with a thoraco-abdominal cushion or a modified lateral cushion, based on measurements from electrical impedance tomography (EIT), gasometric data, and parameters of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or more, with
* moderate or severe acute respiratory distress syndrome (ARDS), and
* indication of prone position

Exclusion Criteria:

* Contra-indication to the prone position: intracranial pressure > 30 mmHg or cerebral perfusion pressure < 60 mmHg; massive haemoptysis needing urgent surgical or radiological treatment; tracheal or thoracic surgery in the last 15 days; facial trauma or surgery in the last 15 days; deep venous thrombosis or pulmonary embolism treated in the last 2 days; unstable bone dislocations of rachis, femur, rib cage, pelvis; mean systolic arterial pressure less than 70 mmHg despite vasopressive therapy and pregnancy
* Severe acute respiratory distress syndrome (ARDS) caused b coronavirus disease 2019 (despite meeting the Berlin criteria for ARDS, their ventilatory mechanics are characterized by nearly normal compliance, something rarely seen in patients with ARDS from other etiologies)
* contraindications for the use of Electrical Impedance Tomography (EIT) such as presence of a cardiac implantable electronic device
* Pulmonary transplantation
* Prone position before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lung recruitment | 1 hour before prone - 2 hours before supine
  Change in ventilation of dorsal regions of lung (%) assessed by electrical impedance tomography

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Martins de de Oliveira, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No